CLINICAL TRIAL: NCT07031583
Title: Impact of Early Versus Delayed Cord Clamping on Oxidative Stress in Neonates With Intrauterine Growth Restriction: A Prospective Comparative Study
Brief Title: Intrauterine Growth Restriction and Intrauterine Fetal Death
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Collaborators: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Ozge Baykan Copuroglu, Asst. Prof., Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KayseriCityHospital
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Intrauterine Growth Restriction (IUGR); Oxidative Stress in Neonates; Umbilical Cord Clamping Time
Keywords: Umbilical Cord Clamping; Fetal Growth Restriction; Oxidative Stress; Total Antioxidant Capacity; Total Oxidant Status
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Four-group parallel design based on neonatal growth status and cord clamping timing.
Who Masked: Outcomes Assessor
Masking Description: The laboratory personnel responsible for analyzing the biochemical markers (TAS, TOS, and catalase) were blinded to the group assignments of the neonates. Samples were coded and processed anonymously to ensure objective assessment of oxidative stress parameters. Other study personnel, including those involved in clinical procedures, were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IUGR-Delayed Cord Clamping (IUGR-DCC) (Experimental): Neonates diagnosed with intrauterine growth restriction (IUGR) received delayed umbilical cord clamping, performed 60-180 seconds after birth. Umbilical cord blood samples were collected immediately for oxidative stress analysis.
  Interventions: Procedure: Delayed Umbilical Cord Clamping (DCC)
- IUGR - Early Cord Clamping (IUGR-ECC) (Active Comparator): Neonates with IUGR underwent early umbilical cord clamping, within 60 seconds after birth. Umbilical cord blood samples were collected for comparison with delayed clamping groups.
  Interventions: Procedure: Early Umbilical Cord Clamping (ECC)
- AGA - Delayed Cord Clamping (AGA-DCC) (Experimental): Neonates appropriate for gestational age (AGA) underwent delayed cord clamping, performed 60-180 seconds after birth. Biochemical markers of oxidative stress were measured using cord blood samples.
  Interventions: Procedure: Delayed Umbilical Cord Clamping (DCC)
- AGA - Early Cord Clamping (AGA-ECC) (Active Comparator): AGA neonates received early umbilical cord clamping, within the first 60 seconds post-delivery. Cord blood was analyzed for oxidative stress markers as a baseline comparator.
  Interventions: Procedure: Early Umbilical Cord Clamping (ECC)

INTERVENTIONS:
Procedure: Delayed Umbilical Cord Clamping (DCC) — The umbilical cord was clamped between 60 and 180 seconds after birth or after the cessation of cord pulsation, in accordance with WHO recommendations. This procedure allows for additional placental transfusion and potential enhancement of neonatal antioxidant capacity.
  Arms: AGA - Delayed Cord Clamping (AGA-DCC); IUGR-Delayed Cord Clamping (IUGR-DCC)
Procedure: Early Umbilical Cord Clamping (ECC) — The umbilical cord was clamped within the first 60 seconds after birth. This represents the standard or traditional approach used for comparison with delayed clamping in terms of oxidative stress outcomes.
  Arms: AGA - Early Cord Clamping (AGA-ECC); IUGR - Early Cord Clamping (IUGR-ECC)

SUMMARY:
This study investigated whether delaying the clamping of the umbilical cord after birth can reduce harmful oxidative stress in newborns, especially in those who did not grow well during pregnancy (intrauterine growth restriction - IUGR). By comparing early and delayed cord clamping in 90 newborns, researchers found that delayed clamping improved antioxidant protection and reduced signs of oxidative damage. These benefits were more significant in babies with IUGR. The results suggest that delaying cord clamping could help support better early health outcomes in vulnerable newborns.

DETAILED DESCRIPTION:
This prospective, randomized clinical study examined the effects of early versus delayed umbilical cord clamping on oxidative stress in newborns, with a specific focus on those diagnosed with intrauterine growth restriction (IUGR). Oxidative stress occurs when the body has an imbalance between harmful molecules (oxidants) and protective defenses (antioxidants), which may negatively affect newborns, especially those who experienced limited growth in the womb.

A total of 90 newborns were included and grouped based on their growth status (IUGR or appropriate for gestational age) and the timing of cord clamping (early: within 60 seconds; delayed: after 60-180 seconds). Blood samples were taken from the umbilical cord immediately after birth to measure markers of oxidative stress and antioxidant activity.

The study found that delayed cord clamping was associated with improved antioxidant levels and reduced oxidative stress, particularly in growth-restricted infants. These findings suggest that delaying cord clamping may provide protective health benefits for high-risk newborns.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at ≥29 weeks of gestation
* Diagnosed with Intrauterine Growth Restriction (IUGR) or classified as Appropriate for Gestational Age (AGA) based on prenatal ultrasonography
* For IUGR group: estimated fetal weight below the 10th percentile and abnormal umbilical artery Doppler findings (e.g., elevated resistance index, absent or reversed end-diastolic flow)
* Neonates delivered at Kayseri City Hospital
* Informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Major congenital anomalies or structural malformations
* Intrauterine infections
* Preterm birth before 29 weeks of gestation
* Fetal hydrops
* Maternal conditions such as preeclampsia, gestational diabetes, or systemic disease
* Emergency cesarean delivery
* Neonates requiring immediate postnatal intubation or invasive resuscitation
* Signs of severe perinatal distress preventing umbilical cord sampling

Ages: 0 Hours to 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Total Antioxidant Status (TAS) | At birth (within 30 minutes postpartum)
  TAS levels in umbilical cord blood will be measured using a validated colorimetric method (Erel, 2004). Higher values indicate greater antioxidant capacity.
Total Oxidant Status (TOS) | At birth (within 30 minutes postpartum)
  TOS levels in umbilical cord blood will be assessed using a spectrophotometric assay (Erel, 2005). Elevated levels reflect greater oxidative stress.
Oxidative Stress Index (OSI) | At birth (within 30 minutes postpartum)
  OSI will be calculated as the ratio of TOS to TAS multiplied by 10. It provides a combined indicator of oxidative balance.

SECONDARY OUTCOMES:
Catalase Enzyme Activity | At birth (within 30 minutes postpartum)
  Catalase activity in umbilical cord blood will be measured via spectrophotometry. Catalase is an endogenous antioxidant enzyme that reflects neonatal oxidative defense capacity.
1-Minute and 5-Minute APGAR Scores | Within 5 minutes after birth
  Clinical scoring system evaluating neonatal adaptation at 1 and 5 minutes of life (heart rate, respiration, muscle tone, reflex, color). Higher scores indicate better clinical condition.
Birth Weight | At birth
  Neonatal birth weight (in grams) will be recorded and compared across groups to evaluate any association with clamping time and oxidative status.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel Ghany EA, Alsharany W, Ali AA, Youness ER, Hussein JS. Anti-oxidant profiles and markers of oxidative stress in preterm neonates. Paediatr Int Child Health. 2016 May;36(2):134-40. doi: 10.1179/2046905515Y.0000000017. PMID 25940692
- [Derived] Demir MB, Copuroglu M, Ozdemir A, Kocer D. Impact of early versus delayed cord clamping on oxidative stress in neonates with intrauterine growth restriction: a prospective randomized controlled trial. BMC Pregnancy Childbirth. 2025 Dec 5;25(1):1291. doi: 10.1186/s12884-025-08335-z. PMID 41350641